CLINICAL TRIAL: NCT01633619
Title: European Implant Cohort Study
Acronym: EICS
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Centre Hospitalier Universitaire Vaudois (Other)
Responsible Party: Principal Investigator, Andrej Trampuz, Medical Doctor, Centre Hospitalier Universitaire Vaudois
Other Study IDs: CHUV0005
Record Dates: First submitted 2012-07-02; First posted 2012-07-04 (Estimated); Last update posted 2012-07-04 (Estimated); Status verified 2012-07

CONDITIONS: Bone Diseases
Keywords: Prosthetic Joint Infection
MeSH Terms: conditions — Bone Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The incidence of postoperative PJI is ranging from 0.5-2.5% for primary interventions and are reported up to 20% for revision procedure. In addition, hematogenous PJI can occur at any time after implantation and the risk of infection remains during the entire prosthesis indwelling time. Prosthetic joint infections (PJI) are associated with significant morbidity and costs to the healthcare system. Evidence for optimal management of PJI with best outcome and lowest expenses is limited and recommendations between countries vary significantly. There is unmet need to standardized diagnostic procedures and definition of infection as well as achieve a consensus for uniform treatment guidelines.The European Implant Cohort Study (EICS) is a multicenter European research project, including patients with PJI in a cohort representative for Europe. The EICS is established jointly by the Orthopedic and Traumatology surgeons, Infectious Diseases specialists and microbiologists of selected university and non-university institutions across Europe. The principal aim of the EICS is to improve the management of PJI and develop consensus guidelines across Europe. By systematic analysis of consecutively included patients with PJI, factors associated with best outcome regarding infection (assessed by the infection-free interval) and joint function (assessed by the degree of pain, mobility, range of motion) will be determined in a longitudinal prospective study with long-term follow-up. This is an investigator-initiated, open, prospective, multicenter observational study. Participating study centers will be university or non-university hospitals across Europe, which fulfill the following study conditions:

* Close collaboration between infectious diseases specialists, microbiologists and orthopedic/trauma surgeons,
* Availability of appropriate microbiological methods (following standard recommendations including sonication of removed prosthesis),
* Availability a dedicated study team (study nurse and/or research fellow) for regular eligibility screenings, patient inclusion procedure, real-time data collection and patient follow-up.

This project may generate important scientific evidence for future guidelines regarding management of PJI, has the potential to initiate new multicenter substudies in an establish network, and may open further collaboration and exchange of skills between institutions across Europe.

DETAILED DESCRIPTION:
INTRODUCTION

1. Objectives

   The principal aim of the EICS is to improve the management of PJI and develop consensus guidelines across Europe. By systematic analysis of consecutively included patients with PJI, factors associated with best outcome regarding infection (assessed by the infection-free interval) and joint function (assessed by the degree of pain, mobility, range of motion) will be determined in a longitudinal prospective study with long-term follow-up.

   In the EICS evaluable patient groups will be generated enabling the comparison between different surgical and antimicrobial treatment concepts. This study aim will be achieved by:

   - Recruitment of patients with PJI of joint prostheses (e.g. hip, knee, shoulder and ankle joints) in participating study centers.
   * Systematic collection of clinical, radiological, pharmacological, laboratory, microbiological, treatment and outcome data using a standardized electronic CRF (eCRF)
   * Ensuring long-term follow-up of patient with evaluation regarding infection, functional result and health care costs.
2. Background

   Orthopedic devices are increasingly used for treatment of the degenerative joint disease and for fixation of bone fractures in the growing population of the elderly. In the United States, about 800,000 primary hip and knee arthroplasties were performed in 2006; by the year 2030, the demand for primary total hip arthroplasties is estimated to increase to 572,000 and for primary total knee arthroplasties to 3.48 million procedures. Similar increase of primary and revision arthroplasty surgeries are observed in Europe.

   Due to high cost of implantable devices and considerably morbidity associated with surgical procedure, a non-invasive approach is the preferred treatment modality, if possible (i.e. retention of the implant with antibiotic therapy active against biofilms).
3. Purpose of the study

The EICS is a multicenter European research project, including patients with prosthetic joint infections (PJI) in a cohort representative for Europe. The European Implant Cohort Study is established jointly by the Orthopedic and Traumatology surgeons, Infectious Diseases specialists and microbiologists of selected university and non-university institutions across Europe.

RESEARCH PLAN

1. Study design

   This is an investigator-initiated, open, prospective, multicenter observational study. Participating study centers will be university or non-university hospitals across Europe, which fulfill the following study conditions:
   * Close collaboration between infectious diseases specialists, microbiologists and orthopedic/trauma surgeons,
   * Availability of appropriate microbiological methods (following standard recommendations including sonication of removed prosthesis),
   * Availability a dedicated study team (study nurse and/or research fellow) for regular eligibility screenings, patient inclusion procedure, real-time data collection and patient follow-up.
2. Material and Methods

   1. Patient recruitment, ethics and study procedure All patients with a suspected PJI will be screened for eligibility by the responsible research fellow in each participating study center. Potential study participants will be identified during the outpatient visit (before hospitalization) or after admission. The data will be collected using an electronic Case Report Form (eCRF) in real-time (within 5 days of patient inclusion). The approval of the Institutional Review Board (IRB) will be obtained before start of the study. Patients will give informed consent before study inclusion. The study protocol will be submitted for evaluation to the European Medicines Agency (EMA). For all local study coordinators a training workshop will be organized before start of recruitment. In addition, a hotline is available for questions regarding the inclusion/exclusion procedure, data collection, treatment algorithm or adverse event reporting.
   2. Data collection The following data will be collected at study inclusion, during hospitalization and during follow-up visits (3, 6, 12 months and thereafter as the usual clinical practice): demographic data, date of primary implantation, type of implant, previous joint surgeries, presence of potential risk factors for PJI, clinical characteristics, microbiological, laboratory and radiological data. At each follow-up visit, functional outcome, adherence to antimicrobial treatment protocol, potential drug-drug interactions and possible side effects of antimicrobials will be recorded. Patients who will not appear at their scheduled visits will be actively contacted by phone (or their treating practitioners).
   3. Outcome evaluation

      The following outcome endpoints will be evaluated:

      • Primary outcome: Infection outcome. This will be determined as the infection-free interval after end of treatment. Infection-free status is defined as absence of clinical (e.g. no fistula), laboratory (e.g. normal C-reactive protein) and radiological signs of infection (e.g. no septic loosening). The expected "cure rate", defined as the infection-free interval at 2 years, is > 80%. The treatment outcome of the combined (antimicrobial and surgical) treatment approach will be assessed in a time-dependent manner using the Kaplan-Meier survival method.
      * Secondary outcome: Functional outcome and pharmacokinetic studies. The functional assessment will be performed using joint-specific scores involving the range of motion (ROM), patient mobility / independency in daily life and subjective evaluation of pain using a pain scale (1-10 points). The expected functional outcome is that >60% patients return to previous life activities, > 75% reduction of pain.

      Definitions of variables

      • If clinical, laboratory or radiographic signs are suggesting infection, preoperative (e.g. arthrocentesis) and/or intraoperative procedures (e.g. arthroscopy or arthrotomy) will be performed to proactively confirm or exclude an infection. In case of uncertainty, diagnostic procedure will be repeated in several days to weeks (depending on the severity of symptoms).

      • PJI is defined if at least one of the following criteria are present: (i) presence of sinus tract (fistula), (ii) increased leukocyte count or neutrophils percentage in preoperative synovial fluid aspirate, (iii) acute inflammation in histopathology of periprosthetic tissue, (iv) visible pus around the prosthesis, (v) growth in synovial fluid, sonication or periprosthetic tissue.
      * Further classification is performed according to the route of infection (intraoperative or hematogenous) and clinical presentation (acute versus chronic = low-grade).
      * Device outcome is evaluated regarding infection (i.e. primary outcome = new infection with a different pathogen versus persistent infection with same organism) or functionality (i.e. secondary outcome = concerning non-infectious characteristics, such as aseptic device failure, periprosthetic or implant fracture, pain, mobility).
      * The number of variables, which will be evaluated with regard to treatment outcome are reduce to the following 3 parameters: (i) type of joint prosthesis, (ii) type of surgical procedure, (iii) type of antimicrobial treatment. If the patient is not treated according to the predetermined treatment protocol (i.e. study protocol deviation), these patients will be evaluated separately.

        d. Microbiology diagnostic Microbiology analyses will be performed at the local microbiology laboratories of each participating study center. The antimicrobial susceptibility of isolated microorganisms will be tested by as routine practice. Synovial fluid will be aspirated preoperatively (when appropriate) and multiple (at least 3 specimens) periprosthetic tissue samples will be collected during initial surgery. All isolated strains will be re-identified and their antimicrobial susceptibility will be re-tested at the central microbiology laboratory. In addition, the explanted prosthesis (or part of it) will be investigated by sonication to increase the diagnostic yield of biofilms by detachment of adherent microorganism.

        e. Pharmacokinetic studies In selected study centers (optional), population pharmacokinetic profile of the administered antimicrobials (e.g. daptomycin, rifampicin, vancomycin) in plasma and in drainage fluid will be determined, to quantify inter- and intra-patient variability and to identify sources of variability in drug concentrations.

        f. Safety Adverse events and Serious Adverse events (SAE)
      * An adverse event is the appearance or worsening of any undesirable sign, symptom, or medical condition occurring after starting study medication even if the event is not considered to be related to study medication. Medical conditions/diseases present before starting study medication are only considered adverse events if they worsen after starting the study medication. Abnormal laboratory values or test results constitute adverse events only if they induce clinical signs or symptoms, are considered clinically significant, or require therapy.
      * An SAE is defined as an event which:

        * Is fatal or life-threatening
        * Results in persistent or significant disability/incapacity
        * Constitutes a congenital anomaly/birth defect
        * Requires inpatient hospitalization or prolongation of existing hospitalization, unless hospitalization is for: routine treatment or monitoring of the studied indication, not associated with any deterioration in condition ; elective or pre-planned treatment for a pre-existing condition that is unrelated to the indication under study and has not worsened since the start of daptomycin ; treatment on an emergency outpatient basis for an event not fulfilling any of the definitions of a SAE given above and not resulting in hospital admission ; social reasons and respite care in the absence of any deterioration in the patient's general condition

          g. Data analysis Depending on the type of data, the results are expressed as mean ± SD or number of subjects (percentage). For each method, the factors that influence the functional status of participants will be identified first by a bivariate survival analysis (Kaplan-Meyer). This first analysis will identify a number of potential risk factors, which will be later confirmed by a multivariate survival analysis (Cox regression model). The results are expressed as relative risk and 95% confidence interval. The success rate at two years of each method is then compared with literature values by a chi-square test.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is older than 18 years of age.
2. Written Informed consent has been obtained.
3. Subject has a prosthetic joint infection (PJI) of the hip, knee or shoulder prosthesis defined as presence of at least one of the following criteria:

   * visible pus around the prosthesis
   * presence of sinus tract (fistula),
   * acute inflammation in histopathology of periprosthetic tissue
   * positive microbiology of synovial fluid, sonication or periprosthetic tissue
   * increased leukocyte count or neutrophil percentage in preoperative synovial fluid aspirate,
4. Subject is willing to participate in the study, to follow protocol study treatment regimen, and to comply with all planned follow-up assessments.

Exclusion Criteria:

1. Subject has been previously enrolled in the study or is currently enrolled in another investigational study, which deviates from the treatment algorithm.
2. Inability to read and understand the participant's information.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patient with hip, knee and shoulder prosthetic joint infection.
Sampling Method: Probability Sample
Enrollment: 4000 (Estimated)
Dates: Start 2013-01; Primary Completion 2015-01 (Estimated)

PRIMARY OUTCOMES:
Infection Outcome | 2 years
  This will be determined as the infection-free interval after end of treatment. Infection-free status is defined as absence of clinical (e.g. no fistula), laboratory (e.g. normal C-reactive protein) and radiological signs of infection (e.g. no septic loosening). The expected "cure rate", defined as the infection-free interval at 2 years, is >80%. The treatment outcome of the combined (antimicrobial and surgical) treatment approach will be assessed in a time-dependent manner using the Kaplan-Meier survival method.

SECONDARY OUTCOMES:
Functional outcome | The following data will be collected at study inclusion, during hospitalization and during follow-up visits (3, 6, 12 months and thereafter as the usual clinical practice):
  The functional assessment will be performed using joint-specific scores involving the range of motion (ROM), patient mobility / independency in daily life and subjective evaluation of pain using a pain scale (1-10 points). The expected functional outcome is that >60% patients return to previous life activities, >75% reduction of pain.

CONTACTS AND LOCATIONS:
Overall Officials: Andrej Trampuz, MD, Principal Investigator — Centre Hospitalier Universitaire Vaudois (CHUV), Lausanne; Olivier Borens, MD, Principal Investigator — Centre Hospitalier Universitaire Vaudois (CHUV), Lausanne
Locations (1):
- Centre Hospitalier Universitaire Vaudois (CHUV), Lausanne, Canton of Vaud, Switzerland

REFERENCES:
- [Background] Zimmerli W, Trampuz A, Ochsner PE. Prosthetic-joint infections. N Engl J Med. 2004 Oct 14;351(16):1645-54. doi: 10.1056/NEJMra040181. No abstract available. PMID 15483283
- [Background] Trampuz A, Hanssen AD, Osmon DR, Mandrekar J, Steckelberg JM, Patel R. Synovial fluid leukocyte count and differential for the diagnosis of prosthetic knee infection. Am J Med. 2004 Oct 15;117(8):556-62. doi: 10.1016/j.amjmed.2004.06.022. PMID 15465503
- [Background] Schinsky MF, Della Valle CJ, Sporer SM, Paprosky WG. Perioperative testing for joint infection in patients undergoing revision total hip arthroplasty. J Bone Joint Surg Am. 2008 Sep;90(9):1869-75. doi: 10.2106/JBJS.G.01255. PMID 18762646
- [Background] Atkins BL, Athanasou N, Deeks JJ, Crook DW, Simpson H, Peto TE, McLardy-Smith P, Berendt AR. Prospective evaluation of criteria for microbiological diagnosis of prosthetic-joint infection at revision arthroplasty. The OSIRIS Collaborative Study Group. J Clin Microbiol. 1998 Oct;36(10):2932-9. doi: 10.1128/JCM.36.10.2932-2939.1998. PMID 9738046
- [Background] Trampuz A, Piper KE, Jacobson MJ, Hanssen AD, Unni KK, Osmon DR, Mandrekar JN, Cockerill FR, Steckelberg JM, Greenleaf JF, Patel R. Sonication of removed hip and knee prostheses for diagnosis of infection. N Engl J Med. 2007 Aug 16;357(7):654-63. doi: 10.1056/NEJMoa061588. PMID 17699815
- [Background] Kurtz SM, Ong KL, Schmier J, Mowat F, Saleh K, Dybvik E, Karrholm J, Garellick G, Havelin LI, Furnes O, Malchau H, Lau E. Future clinical and economic impact of revision total hip and knee arthroplasty. J Bone Joint Surg Am. 2007 Oct;89 Suppl 3:144-51. doi: 10.2106/JBJS.G.00587. No abstract available. PMID 17908880